CLINICAL TRIAL: NCT02097407
Title: Preoperative Dexmedetomidine Reduces the EC50 of Propofol for Successful i-gelTM Insertion Without Muscle Relaxants
Brief Title: Preoperative Dexmedetomidine & EC50 of Propofol
Acronym: PreopDXM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Pyoung Park, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PreopDXM_PPF
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Urologic Surgery

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group D : Dexmedetomidine + propofol group (Experimental): In Group D, DEX (1 µg kg-1) was intravenously loaded for 10 min before induction of anaesthesia.
  Interventions: Drug: Group D : Dexmedetomidine + propofol group
- Group C : Saline + propofol group (Placebo Comparator): In Group C, 0.9% of normal saline (1 µg kg-1) was loaded 10 min before induction of anaeshtesia.
  Interventions: Drug: Group C : Saline + propofol group

INTERVENTIONS:
Drug: Group C : Saline + propofol group — All patients were pre-oxygenated with 100% oxygen with spontaneous breathing for 3 min before the end of loading of normal saline. Anaesthesia was induced with predetermined effect-site propofol concentrations using a target-controlled infusion device (Orchestra; Fresenius-Vial, Brezins, France). The first patient in Group C received an effect-site propofol concentration of 3 and 5 µg mL-1, respectively, over 5 min.
  After equilibration of the plasma and effect-site propofol concentrations, i-gel (size 4 for patients weighing 50-90 kg, size 3 for patients weighing 30-50 kg) was inserted using the standard technique by a single anaesthesiologist staff member with expertise in i-gel insertion and who entered the operating room immediately before i-gel insertion to blind him to the group assignment
  Arms: Group C : Saline + propofol group
Drug: Group D : Dexmedetomidine + propofol group — All patients were pre-oxygenated with 100% oxygen with spontaneous breathing for 3 min before the end of loading of dexmedetomidine. Anaesthesia was induced with predetermined effect-site propofol concentrations using a target-controlled infusion device (Orchestra; Fresenius-Vial, Brezins, France). The first patient in Group D received an effect-site propofol concentration of 3 and 5 µg mL-1, respectively, over 5 min.
  After equilibration of the plasma and effect-site propofol concentrations, i-gel (size 4 for patients weighing 50-90 kg, size 3 for patients weighing 30-50 kg) was inserted using the standard technique by a single anaesthesiologist staff member with expertise in i-gel insertion and who entered the operating room immediately before i-gel insertion to blind him to the group assignment.
  Arms: Group D : Dexmedetomidine + propofol group

SUMMARY:
Dexmedetomidine is a useful anaesthetic adjuvant for general anaesthesia. In this prospective randomised study, we determined whether preoperative dexmedetomidine administration could reduce the half maximal effective concentration (EC50) of propofol for successful i-gelTM insertion without muscle relaxants.

DETAILED DESCRIPTION:
Propofol is a useful induction agent for LMA insertion without muscle relaxants because it profoundly inhibits pharyngeal and laryngeal reactivity. A previous report showed that the effect-site concentration of propofol for successful classic LMA insertion in 50% of adults (EC50) without muscle relaxants in healthy male patients was 8.72 (0.55) µg ml-1. The EC50 of propofol may be dependent on the type of LMA used. A previous study comparing the EC50 of the propofol concentration between classic and proseal LMA insertions demonstrated that the EC50 of propofol needed for proseal LMA insertion was 35% greater than that needed for classic LMA insertion. Unfortunately, no investigation has been performed to determine the EC50 of the propofol concentration required for i-gel insertion without muscle relaxants.

Dexmedetomidine (DEX), a selective alpha-2 agonist, has sympatholytic, sedative, and analgesic properties. Such beneficial characteristics make DEX a useful anaesthetic adjuvant for general anaesthesia. Many reports have revealed the beneficial effects of DEX in terms of reducing intraoperative anaesthetic requirements, postoperative analgesic demand, and increased haemodynamic responses to noxious stimuli such as endotracheal intubation. A previous investigation showed that preoperative clonidine, an alpha-2 agonist, decreased the EC50 required for LMA insertion.

We hypothesised that preoperative DEX administration can reduce the propofol concentration required for i-gel insertion. In this study, we compared the EC50 of propofol needed for successful i-gel insertion without muscle relaxants between DEX and placebo groups

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients who were 20-65 years old and scheduled for general anaesthesia for urologic surgery

Exclusion Criteria:

* Patients with an allergy to alpha-2 adrenergic agonists or propofol
* Patients who anticipated difficult airway (cervical spinal disease, Mallampati score of III or IV, a mouth opening of <2.5 cm, and/or body mass index of >30 kg m-2), unstable teeth
* Patients with bradycardia of <50 beats/min, heart block greater than first degree, severe cardiorespiratory dysfunction
* Patients with symptoms of upper respiratory infection

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
EC50 of propofol required for successful i-gel insertion | During i-gel insertion anticipated up to 1 min
  The EC50 of propofol for successful i-gel insertion was determined by a modification of Dixon's up-and-down method. The response of each patient determined the effect-site propofol concentration for the next patient. If the response was deemed 'successful', the next target concentration of propofol was decreased by 0.5 µg mL-1. If the response was deemed a 'failure', the target concentration was increased by the same dose. The process was repeated until the sixth crossover point (success/failure) was obtained.

SECONDARY OUTCOMES:
the total dose of propofol infused before i-gel insertion | During i-gel insertion time anticipated upto 1min
  The total amount of propofol infused before i-gel insertion was noted. The insertion time, defined as the time from picking up the i-gel until the initiation of mechanical ventilation.
the presence/severity of airway trauma after i-gel insertion | At the time point of removing the i-gel from patient's mouth
  After removing the i-gel, airway trauma (defined as any blood staining on the device) was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Pyung Park, MD PhD, Study Director — Professor; Young Cheol Kim, Md PhD, Principal Investigator — Professor
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jang YE, Kim YC, Yoon HK, Jeon YT, Hwang JW, Kim E, Park HP. A randomized controlled trial of the effect of preoperative dexmedetomidine on the half maximal effective concentration of propofol for successful i-gel insertion without muscle relaxants. J Anesth. 2015 Jun;29(3):338-345. doi: 10.1007/s00540-014-1949-9. Epub 2014 Nov 14. PMID 25394762